CLINICAL TRIAL: NCT04340518
Title: Measuring the Recovery of the Conjunctival Tissue After 4 Days of Scleral Lens Wear
Brief Title: Conjunctival Rebound After Scleral Lens Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, MKWalker, Instructor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00001908
Record Dates: First submitted 2020-02-03; First posted 2020-04-09 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Conjunctival Diseases
Keywords: scleral lenses
MeSH Terms: conditions — Conjunctival Diseases

STUDY DESIGN:
Intervention Model Description: Prospective observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Post-scleral lens wear (Experimental): Normal subjects without ocular diseased who have worn scleral lenses for at least 8 hours.
  Interventions: Device: Scleral lens

INTERVENTIONS:
Device: Scleral lens — Scleral contact lenses, manufactured in rigid gas permeable fluorosilicone acrylate polymers and treated with plasma treatment prior to use.

SUMMARY:
Scleral lenses, customized rigid contact lenses that land on the soft and spongy conjunctival tissue overlying the sclera, will be fitted on 15 subjects with normal ocular surfaces. The purpose of the study is to determine the amount of conjunctival compression caused by the devices and the length of time required for the shape to recover from compression.

DETAILED DESCRIPTION:
The purpose of this study is to determine the interval required for the conjunctival tissue to return to its natural shape after scleral lens wear. All study visits will take place at the University of Houston College of Optometry (UHCO). Subjects will be recruited and fitted with scleral lenses to wear during the experimental days. Once the proper fit has been achieved, subjects will wear the scleral lens for 4 days total, returning after the 1st and 4th day of lens wear for approximately 2 hours of testing. The subjects will then return every 24-hours for measurements until their conjunctival shape has returned to the original shape. The testing will be done using the sMap scleral topographer, which measures the elevation of the conjunctiva. Testing is non-invasive although it requires instillation of Fluress eye drops, a sodium fluorescein dye with anesthetic that allows for imaging. The total number of visits is 9-14 and the length of visit ranges from 10 minutes to 2.5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Normal ocular surface without conjunctival or scleral disease
* Male or female
* 18 years of age and older prior to the initial visit
* A non-scleral lens wearer.

Exclusion Criteria:

* Individuals with anterior segment ocular pathology that may affect intraocular pressure and/or scleral/conjunctival health.
* Individuals with known adverse response to Fluress® ophthalmic drops
* Individuals with a history of habitual scleral lens wear
* If a usable baseline image is unable to be obtained at the initial visit due to small ocular surface area or eyelid anatomy
* Individuals currently taking any ocular medications that could affect intraocular pressure and/or scleral/conjunctival health
* Individuals who have any other conditions or situations which, in the investigator's opinion, may put the subject at significant risk, may confound study outcomes, or may significantly interfere with the subject's participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Rebound at 120 minutes post-SL removal, Day 4 | Measured 120-130 minutes post-SL removal, Day 4
  Conjunctival rebound amount at 120 minutes post-removal, Day 4

SECONDARY OUTCOMES:
Rebound at 120-hours post-SL discontinuation | Measured 115-125 hours post-SL removal
  Conjunctival rebound amount at 120 hours post-removal
Rebound at 168-hours post-SL discontinuation | Measured 160-170 hours post-SL removal
  Conjunctival rebound amount at 168 hours post-removal
Rebound at 144-hours post-SL discontinuation | Measured 140-150 hours post-SL removal
  Conjunctival rebound amount at 144 hours post-removal
Rebound at 72-hours post-SL discontinuation | Measured 60-80 hours post-SL removal
  Conjunctival rebound amount at 72 hours post-removal
Rebound at 90 minutes post-SL removal, Day 4 | Measured 90-100 minutes post-SL removal, Day 4
  Conjunctival rebound amount at 90 minutes post-removal, Day 4
Rebound at 90 minutes post-SL removal, Day 1 | Measured 90-100 minutes post-SL removal, Day 1
  Conjunctival rebound amount at 90 minutes post-removal, Day 1
Rebound at 60 minutes post-SL removal, Day 4 | Measured 60-70 minutes post-SL removal, Day 4
  Conjunctival rebound amount at 60 minutes post-removal, Day 4
Rebound at 30 minutes post-SL removal, Day 1 | Measured 30-40 minutes post-SL removal, Day 1
  Conjunctival rebound amount at 30 minutes post-removal, Day 1
Rebound at 24-hours post-SL discontinuation | Measured 20-30 hours post-SL removal
  Conjunctival rebound amount at 24 hours post-removal
Rebound at 5 minutes post-SL removal, Day 1 | Measured 5-10 minutes post-SL removal, Day 1
  Conjunctival rebound amount at 5 minutes post-removal, Day 1
Rebound at 30 minutes post-SL removal, Day 4 | Measured 30-40 minutes post-SL removal, Day 4
  Conjunctival rebound amount at 30 minutes post-removal, Day 4
Rebound at 120 minutes post-SL removal, Day 1 | Measured 120-130 minutes post-SL removal, Day 1
  Conjunctival rebound amount at 120 minutes post-removal, Day 1
Rebound at 5 minutes post-SL removal, Day 4 | Measured 5-10 minutes post-SL removal, Day 4
  Conjunctival rebound amount at 5 minutes post-removal, Day 4
Rebound at 60 minutes post-SL removal, Day 1 | Measured 60-70 minutes post-SL removal, Day 1
  Conjunctival rebound amount at 60 minutes post-removal, Day 1
Rebound at 48-hours post-SL discontinuation | Measured 40-50 hours post-SL removal
  Conjunctival rebound amount at 48 hours post-removal
Rebound at 96-hours post-SL discontinuation | Measured 90-100 hours post-SL removal
  Conjunctival rebound amount at 96 hours post-removal

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston College of Optometry, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided